CLINICAL TRIAL: NCT05346224
Title: A Multicenter, Randomized, Double-Blind, Parallel-Controlled Phase III Clinical Study to Evaluate the Efficacy and Safety of Pertuzumab Biosimilar HLX11 vs. EU-Perjeta® in the Neoadjuvant Therapy of HER2-Positive and HR-Negative Early-stage or Locally Advanced Breast Cancer
Brief Title: A Study to Evaluate the Efficacy and Safety of HLX11 vs. EU-Perjeta® in the Neoadjuvant Therapy of HER2-Positive and HR-Negative Early-stage or Locally Advanced Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX11-BC301
Record Dates: First submitted 2022-04-17; First posted 2022-04-26 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Breast Neoplasms; HER2-positive Breast Cancer
Keywords: Perjeta; Pertuzumab; early-stage; locally Advanced; neoadjuvant; adjuvant
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Parallel-Controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment group (Experimental): HLX11 combined with trastuzumab and docetaxel will be adopted in the neoadjuvant treatment phase, and doxorubicin with cyclophosphamide will be administered in the adjuvant chemotherapy treatment phase, HLX11 combined with trastuzumab will be administered in the adjuvant treatment phase for HER-2 targeted.
  Interventions: Drug: HLX11
- Control group (Active Comparator): Perjeta combined with trastuzumab and docetaxel will be adopted in the neoadjuvant treatment phase, and doxorubicin with cyclophosphamide will be administered in the adjuvant chemotherapy treatment phase, HLX11 or Perjeta combined with trastuzumab will be administered in the adjuvant treatment phase for HER-2 targeted.
  Interventions: Drug: EU-Perjeta®

INTERVENTIONS:
Drug: HLX11 — Neoadjuvant(q3w/cycle，total 4cycle): HLX11(loading dose of 840 mg IV , followed by 420 mg IV q3w)+trastuzumab(loading dose of 8 mg/kg IV, followed by 6mg/kg IV q3w)+docetaxel(75mg/m2 IV q3w) Adjuvant: doxorubicin( 60 mg/m2 IV q3w)+cyclophosphamide( 600 mg/m2 IV q3w),total 4 cycle; trastuzumab(loading dose of 8mg/m2 IV , followed by 6 mg/m2 IV q3w)+HLX11(loading dose of 840 mg IV , followed by 420 mg IV q3w), 13cycle
  Other Names: Recombinant anti-HER2 domain II humanized monoclonal antibody injection
  Arms: Treatment group
Drug: EU-Perjeta® — Neoadjuvant(q3w/cycle，total 4cycle): Perjeta (loading dose of 840 mg IV , followed by 420 mg IV q3w)+trastuzumab(loading dose of 8 mg/kg IV, followed by 6mg/kg IV q3w)+docetaxel(75mg/m2 IV q3w) Adjuvant: doxorubicin( 60 mg/m2 IV q3w)+cyclophosphamide( 600 mg/m2 IV q3w),total 4 cycle; trastuzumab(loading dose of 8mg/m2 IV , followed by 6 mg/m2 IV q3w)+HLX11 or Perjeta (loading dose of 840 mg IV , followed by 420 mg IV q3w), 13cycle
  Arms: Control group

SUMMARY:
This is a phase III, double-blind, randomized, parallel-controlled, multicenter equivalence study to compare the efficacy and safety of pertuzumab biosimilar HLX11 vs. EU-Perjeta® on HER2-positive and HR-negative early-stage or locally advanced breast cancer with a primary tumor > 2 cm.

Patients are random assignment to 2 arms and treatment with either HLX11 or EU-Perjeta® , and received neoadjuvant THP regimen every 3- weeks 4 cycles，adjuvant AC every 3- weeks 4 cycles and pertuzumab+trastuzumab(HP) every 3- weeks 13cycles.

DETAILED DESCRIPTION:
This is a phase III, double-blind, randomized, parallel-controlled, multicenter equivalence study to compare the efficacy and safety of pertuzumab biosimilar HLX11 vs. EU-Perjeta® on HER2-positive and HR-negative early-stage or locally advanced breast cancer with a primary tumor > 2 cm.Subjects will be randomly assigned to treatment group (HLX11) or control group (EU-Perjeta®) at 1:1 ratio. The stratification factors include disease category (early-stage vs. locally advanced) and geographic region (Asia vs. non-Asia).

Study drugs will be administered intravenously on a 3-weekly schedule and given consecutively on the same day in the following sequence trastuzumab, followed by pertuzumab and docetaxel(THP regimen) for neoadjuvant，Doxorubicin in combination with cyclophosphamide (AC) for adjuvant chemotherapy, then HP regimen for adjuvant HER2-targeted.

The primary endpoint is total pCR (tpCR) . Secondary efficacy endpoints include breast pCR (bpCR), objective response rate (ORR),Event-free survival (EFS) and Disease-free survival (DFS).

The safety indicators is incidence, type, severity, and causality of all adverse events (including serious adverse events and AESI) based on NCI CTCAE v5.0; Vital signs, physical examination, laboratory tests, cardiac function test, etc.

pharmacokinetic(PK) and immunogenicity is also assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Primary breast cancer that is:

1. Histologically confirmed invasive breast carcinoma with a primary tumor size of > 2 cm by standard local assessment technique;
2. Breast cancer staging ( in accordance with the American Joint Commitee on Cancer(AJCC) staging system (8th edition)): early-stage (T2-3, N0-1, M0) or locally advanced (T2-3, N2 or N3, M0; T4, any N, M0);
3. HER2 positive confirmed by central laboratory, defined as immunohistochemistry (IHC) 3 +, or IHC 2+ and In Situ Hybridization (ISH) positive;
4. Hormone receptor (HR, including estrogen receptor [ER] and progestin receptor [PR]) negative by central laboratory; ER negative is defined as < 1% nuclear staining, and PR negative is defined as < 1% nuclear staining.

2. Left ventricular ejection fraction (LVEF) at baseline (within 42 days prior to randomization) ≥ 55% measured by echocardiography (ECHO) or multiple gated acquisition (MUGA) scan.

3. Adequate major organ function, meeting the following criteria: Hematology (neither blood transfusion nor correction with hematopoietic stimulating factors within 14 days prior to randomization): white blood cell count ≥ 3.0 × 109/L; absolute neutrophil count ≥ 1.5 × 109/L; hemoglobin ≥ 90 g/L; platelet count ≥ 100 × 109/L; Serum chemistry: Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN), total bilirubin ≤ 1.5 × ULN; for subjects with known Gilbert syndrome, total bilirubin ≤ 2 × ULN; alkaline phosphatase ≤ 2.5 × ULN, serum creatinine ≤ 1.5 × ULN.

4. Women of child-bearing potential have a negative result of serum pregnancy test at screening (within 7 days prior to randomization) and not in lactation, or are infertile. Male participants and women of childbearing potential use a "highly effective" contraceptive measures until 7 months after the last dose of investigational/reference product.

Exclusion Criteria:

1. Inflammatory breast cancer.
2. Stage IV (metastatic) breast cancer, bilateral breast cancer, or multicentric (multiple tumors involving more than 1 quadrant) breast cancer.
3. History of other malignancy within 5 years prior to screening (except for who have received radical treatment of carcinoma in situ of the cervix, basal cell carcinoma or squamous cell carcinoma of the skin ).
4. With serious heart disease or medical history, including but not limited to the following conditions:

1) History of documented heart failure or systolic dysfunction with any NYHA classification(LVEF < 50%); 2) High-risk uncontrolled arrhythmia, such as atrial tachycardia with a heart rate> 100 bpm at rest, significant ventricular arrhythmia (e.g.,ventricular tachycardia), or higher-grade atrioventricular (AV) block (i.e.,Mobitz II second-degree AV block or third degree AV block); 3) Unstable angina pectoris, or angina pectoris requiring anti-angina medication; 4) Evidence of transmural myocardial infarction on ECG; 5) Clinically-significant valvular heart disease; 6) Poorly controlled hypertension (systolic blood pressure> 150 mmHg and/or diastolic blood pressure> 100 mmHg).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2022-04-25 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
The total pathological complete response (tpCR) rate assessed by the Independent Review Committee (IRC) | immediately after the surgery
  tpCR is defined as the histological evidence of no malignancy of lymph nodes in the regions of primary lesion and metastasis of breast cancer (i.e., ypT0/is, ypN0 in accordance with the AJCC staging system)

SECONDARY OUTCOMES:
Breast pathologic complete response (bpCR) rate | immediately after the surgery
  bpCR is defined as the histological evidence of no malignancy in the primary lesion of breast cancer, or only carcinoma in situ (i.e., ypT0/Tis in the AJCC staging system, 8th edition)

CONTACTS AND LOCATIONS:
Locations (79):
- China (75):
  - the First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - The first affiliated hospital of Anhui Medical University, Hefei, Anhui
  - The first affiliated hospital of USTC (Anhui Provincial Hospital), Hefei, Anhui
  - Lu'an people's hospital of Anhui ProvinceLuan, Lu'an, Anhui
  - Maanshan People's Hospital, Ma’anshan, Anhui
  - Yijishan Hospital of Wannan Medical College, Wuhu, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - he First Affiliated Hospital of Chongqing Medical University, Chongqi, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou, Guangdong
  - Sun Yat-Sun Yat-sen Hospital affiliated to Sun Yat-sen Universitysen Hospital affiliated to Sun Yat-sen University, Guanzhou, Guangdong
  - Jieyang People's Hospital, Jieyang, Guangdong
  - Meizhou People's Hospital, Meizhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Shantou Central Hospital, Shantou, Guangdong
  - Yue Bei People's Hospital, Shaoguan, Guangdong
  - Affiliated Hospital of Guangdong Medical University, Zhanjiang, Guangdong
  - Zhongshan People's Hospital, Zhongshan, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Affiliated Tumor Hospital of Guizhou Medical University, Guiyang, Guzhou
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Cangzhou Central Hospital, Cangzhou, Hebei
  - Tangshan People's Hospital, Tangshan, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Anyang Cancer Hospital, Anyang, Henan
  - The First Affiliated Hospital of Henan University of science and Technology, Luoyang, Henan
  - Nanyang Central Hospital, Nanyang, Henan
  - The First Affiliated Hospital of the Xinxiang Medical University, Xinxiang, Henan
  - Xinxiang Central Hospital, Xinxiang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital, Tongji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Xiangya Hospital Of Central South University, Changsha, Hunan
  - The Second Xiangya Hospital Of Central South University, Changsha, Hunan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Jiangsu Cancer Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital With Nanjing Medical University, Nanjing, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - affiliated Hospital of Jiangnan University, Wuxi, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Nanchang Third Hospital, Nanchang, Jiangxi
  - The first hospital of Jilin University, Changchun, JIilin
  - The second hospital of dalian medical university, Dalian, Liaoning
  - Liaoning Cancer Hospital & Institute, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shangdong
  - Liaocheng People's Hospital, Liaocheng, Shangdong
  - he Affiliated Hospital of Qingdao University, Qingdao, Shangdong
  - Qingdao Central Hospital, Qingdao, Shangdong
  - Weifang People's Hospital, Weifang, Shangdong
  - Weifang Hospital of traditional Chinese Medicine, Weifang, Shangdong
  - Weihai Municipal Hospital, Weihai, Shangdong
  - Yantai Yuhuangding Hospital, Yantai, Shangdong
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - The First Affiliated Hospital of Xi'an JiaoTong University, Xian, Shanxi
  - Shaanxi Provincial People's Hospital, Xi’an, Shanxi
  - Yuncheng Central Hospital, Yuncheng, Shanxi
  - Sichuan Provincial People's Hospital, Chengdu, Sichuang
  - People's hospital of Deyang city, Deyang, Sichuang
  - Mianyang Central Hospital, Mianyang, Sichuang
  - The second people's hospital of neijiang, Neijiang, Sichuang
  - The second people's hospital of Yibin, Yibin, Sichuang
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital Zhejiang University School Of Medicine, Hangzhou, Zhejiang
  - The Second Affiliated Hospital Zhejiang University School Of Medicine, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
- University of Pécs, Department of Oncotherapy, Pécs, Baranya, Hungary
- Instytut Centrum Zdrowia Matki Polki, Lodz, Łódź Voivodeship, Poland
- Spain (2):
  - Hospital Clínico Universitario de Santiago de Compostela (CHUS), Santiago de Compostela, A Coruna
  - Hospital Arnau de Vilanova de Lleida, Barcelona, Catalonia

REFERENCES:
- [Result] Yang J, Lin L, Long Q, Zhang Q, Sun G, Zhou L, Wang Q, Zhu J, Li F, Hu W. HLX11, a Proposed Pertuzumab Biosimilar: Pharmacokinetics, Immunogenicity, and Safety Profiles Compared to Three Reference Biologic Products (US-, EU-, and CN-Approved Pertuzumab) Administered to Healthy Male Subjects. BioDrugs. 2022 May;36(3):393-409. doi: 10.1007/s40259-022-00534-w. Epub 2022 May 20. PMID 35594017
- See also: Results from this study demonstrated the bioequivalence between HLX11 and US-, EU-, and CN-pertuzumab, supporting further investigation of HLX11 in clinical studies — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC9148872/